CLINICAL TRIAL: NCT05653453
Title: Clinical Study of Tumor Treating Fields Combined with Gemcitabine and Albumin-bound Paclitaxel in the First-line Treatment of Locally Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Healthy Life Innovation Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100-LAPC1
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tumor treating fields combined with Gemcitabine hydrochloride and albumin binding paclitaxel (Experimental): Device: Tumor treating fields Subjects will use tumor treating fields each day
  Drug: Gemcitabine hydrochloride and albumin binding paclitaxel 28 days is a cycle. On the 1st, 8th and 15th days of each cycle, 125 mg/m2 albumin binding paclitaxel will be administered intravenously，1000 mg/m2 gemcitabine hydrochloride will be administered immediately after the infusion of albumin binding paclitaxel.
  Interventions: Device: Tumor treating fields combined with Gemcitabine hydrochloride and albumin binding paclitaxel; Drug: Gemcitabine hydrochloride and albumin binding paclitaxel
- Gemcitabine hydrochloride and albumin binding paclitaxel (Active Comparator): Drug: Gemcitabine hydrochloride and albumin binding paclitaxel 28 days is a cycle. On the 1st, 8th and 15th days of each cycle, 125 mg/m2 albumin binding paclitaxel will be administered intravenously，1000 mg/m2 gemcitabine hydrochloride will be administered immediately after the infusion of albumin binding paclitaxel.
  Interventions: Drug: Gemcitabine hydrochloride and albumin binding paclitaxel

INTERVENTIONS:
Device: Tumor treating fields combined with Gemcitabine hydrochloride and albumin binding paclitaxel — Device: Tumor treating fields Subjects will use tumor treating fields until disease progression or for a maximum of 30 months.
  Drug: Gemcitabine hydrochloride and albumin binding paclitaxel Subjects will receive Gemcitabine hydrochloride and albumin binding paclitaxel until disease progression or for a maximum of 30 months.
  Arms: Tumor treating fields combined with Gemcitabine hydrochloride and albumin binding paclitaxel
Drug: Gemcitabine hydrochloride and albumin binding paclitaxel — Drug: Gemcitabine hydrochloride and albumin binding paclitaxel Subjects will receive Gemcitabine hydrochloride and albumin binding paclitaxel until disease progression or for a maximum of 30 months.

SUMMARY:
The Objectives of this clinical trial is to evaluate the efficacy and safety of tumor treating fields combined with gemcitabine and albumin bound paclitaxel in the treatment of locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 75 (including 18 and 75) of both genders;
2. Expected survival time ≥3 months;
3. Pancreatic adenocarcinoma confirmed by histology/cytology;
4. Locally advanced lesions meeting any of the following criteria without distant metastasis: ① Pancreatic head and neck tumors: a. The tumor invaded the Superior Mesenteric Artery (SMA) more than 180°; b. The tumor invaded the celiac trunk more than 180°; c. Unresectable reconstruction of superior mesenteric vein or portal vein due to tumor invasion or embolism (tumor thrombus or thrombus); d. The tumor extensively invaded the distal jejunal drainage branch of the superior mesenteric vein. ② Pancreatic body/tail tumor: a. The tumor invaded the superior mesenteric artery or celiac trunk more than 180°; b. Celiac trunk and abdominal aorta involvement; c. The superior mesenteric vein or portal vein cannot be resected and reconstructed due to tumor invasion or embolism (tumor thrombus or thrombus).
5. At least one measurable lesion according to revised RECIST version 1.1;
6. ECOG score 0-1;
7. Be able to receive gemcitabine for injection and paclitaxel for injection (albumin-bound) combined therapy according to medical advice;
8. Able to operate tumor treating fields independently or with the help of nursing staff;
9. AE should be restored to normal or CTCAE1 grade after previous treatment;
10. The serum pregnancy test results of female subjects of reproductive age were negative. Female subjects of reproductive age agree to use effective contraception (e.g. hormonal or barrier methods or abstinence) during the study period and for 6 months after the last dose of chemotherapy drugs;
11. Male subjects agree to use effective birth control (such as barrier method or abstinence) and not to donate sperm during the study and within 3 months after the last chemotherapy drug administration;
12. Voluntarily sign the informed consent.

Exclusion Criteria:

1. The subjects has previously received first-line treatment for pancreatic adenocarcinoma;
2. Subjects with contraindications to treatment with gemcitabine for injection and/or paclitaxel for injection (albumin-bound) or known severe allergies to gemcitabine for injection and/or paclitaxel for injection (albumin-bound);
3. Patients had cancer requiring other antitumor therapy within 2 years before enrollment, excluding treated stage I prostate cancer, cervical cancer in situ, breast cancer in situ, and non-melanoma skin cancer;
4. Abnormal bone marrow, heart, liver and kidney function: a. Neutrophil count < 1.5 × 10^9/L, platelet count < 100 × 10^9/L, hemoglobin < 90g/L; The use of blood transfusion, platelet transfusion and erythropoietin was prohibited within 14 days before C1D1, and the use of Leukocytotropic drug such as G-CSF, fegrasstim, pefegrasstim, etc., was prohibited within 7 days before C1D1.b. Total bilirubin > 1.5× Upper Limit of Normal (ULN); Subjects with a total bilirubin > 2×ULN that is elevated due to pancreatic cancer compression of the bile duct but has been fitted with a bile duct stent for drainage can be enrolled. AST and/or ALT> 2.5×ULN; the use of drugs that improve liver function, such as reducing transaminase was prohibited within 7 days before C1D1. c. Serum creatinine > 1.5×ULN; d. A history of severe cardiovascular disease, including but not limited to second or third degree heart block; Severe ischemic heart disease; New York Heart Association (NYHA) class II or higher congestive heart failure (mild physical activity limitation; Comfortable at rest, but normal activities can cause fatigue, palpitations, or difficulty breathing);
5. Subjects who were required to receive systemic corticosteroids (doses equivalent to > 10 mg prednisone/day) or other immunosuppressive agents within 14 days before enrollment or during the study period. Subjects were eligible for enrollment if: a. The use of topical or inhaled glucocorticoids is permitted; b. Allow short-term (≤7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases;
6. Those who had severe infection before the first dose were judged ineligible for the study by the investigator;
7. History of human immunodeficiency virus (HIV) infection (known HIV1/2 antibody positive);
8. The presence of active hepatitis B, active hepatitis C, or other active infections that may affect the patient's treatment as determined by the investigator;
9. Subjects with a clear history of neurological or psychiatric disorders, such as epilepsy, dementia, or substance abuse (including alcohol) within the last year, and possibly affecting compliance;
10. Infected, ulcerated or unhealed wounds exist on the skin where the tumor treating fields is applied;
11. Having an implantable electronic medical device, such as a pacemaker;
12. Metal medical instruments are implanted in the chest and abdomen such as bone nails;
13. Known allergies to medical adhesives or hydrogels;
14. Pregnant or breastfeeding;
15. Subjects participated in clinical trials of other drugs within 3 months before enrollment, or participated in clinical trials of other devices within 1 month before enrollment;
16. Subjects with poor compliance or other factors as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 12 months after the last study treatment
  From date of enrollment until the date of death from any cause

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | The whole study period
  Adverse events will be defined as the incidence, frequency and severity of adverse events (AEs) noted in patients treated with study treatments
Progression-free survival (PFS) | up to 30 months
  Progression-free survival is defined as the time from the start of treatment with Tumor Treating Fields and Docetaxel until the first documentation of disease progression or death due to any cause, whichever occurs first
12-month OS rate | 12 months
  12-month Overall survival rate
Progression Free Survival rate at 6 months | 6 months
  The analysis will be estimated proportions of patients who are progression-free at 6 months based on the RECIST 1.1 criteria following the time of enrollment

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Affiliated Huashan Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality